CLINICAL TRIAL: NCT03952910
Title: An Online Pain Education Program for Working Adults: a Pilot Randomized Controlled Trial With One-month Follow-up
Brief Title: An Online Pain Education Program for Working Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSE Mun Yee Mimi, Associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OPEP
Record Dates: First submitted 2019-05-04; First posted 2019-05-16 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Working adults; Pain education; Internet-delivered
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Online pain education program will be accessible by the intervention group
  Interventions: Other: Online pain education program
- Control group (No Intervention): No intervention for the control group, only one-page simple material related to pain will be provided.

INTERVENTIONS:
Other: Online pain education program — Online pain education program
  Arms: Experimental group

SUMMARY:
Pain is popular among working population and it is a strong predictor of poor quality of life. In this study, an internet-delivered pain education program will be provided to working adults aims at helping patients equip with pain-related knowledge and useful skills and evaluate the effectiveness of the internet-delivered program. Participants will be recruited follow snowball sampling and will be randomly allocated to experimental group and control group by 1:1 ratio. The internet-delivered pain education will last for 4 weeks with one-month follow-up. Basic knowledge of pain, pharmacological and non-pharmacological treatment and related resources will be introduced in the program. Pain intensity, pain-related disability, anxiety, depression and self-efficacy will be measured in baseline post-treatment and at one-month follow-up. Acceptability and satisfaction to the program will also collected.

DETAILED DESCRIPTION:
Participants' eligibility will be accessed based on the following details:

1. Inclusion criteria:

1. . Age between 16 to 60;
2. . Have a full-time job;
3. . Resident of China;
4. . Can read and understand Chinese;
5. . History with non-cancer pain in past 6 months(Nicholas et al., 2013);
6. . Pain score should be at least 2 when using Numeric Rating Scale, a 11-point numeric scale (Pieh et al., 2012);
7. . Own a mobile phone and can access to mobile phone, computer and the internet.

2. Exclusion criteria

1. . Hospitalized patients;
2. . Experiencing a drug addiction problem;
3. . Further medical and surgical treatments or interventions is planned.

The outcome measures will be considered in four aspects, physical, psychological, psycho-social using a battery of questionnaires which were used in the previous similar studies and evaluation to the program will be measured by asking several questions. As the study will be conducted in China, all the questionnaires will use Chinese version.

1. Physical Brief Pain Inventory (BPI): The BPI is a brief, self-administered questionnaire us. Pain severity is assessed by four items and pain interference by seven items. The items are rated on a scale ranging from 0 to 10. Previous study showed that BPI can used to measure not only cancer pain but also chronic pain and proved that BPI has good internal consistency and acceptable test-retest reliability.
2. Psychological Depression Anxiety Stress Scales (DASS): The DASS is a self-report instrument to measure three negative emotional states including depression, anxiety and stress. The previous study demonstrated that DASS has excellent internal consistency and validity was also proved.
3. Psycho-social The Pain Self-efficacy Questionnaire (PSEQ): A 10 item questionnaire assess the patient's beliefs about his or her ability to accomplish daily activities with pain. Higher score indicate greater pain-related self-efficacy.
4. Satisfaction and acceptability Several questions will be asked at the end of the program to assess participants' satisfaction and acceptability of the program: (1) "Do you think this online pain management program useful?" "Does it worth your time following the program?" "Would you feel confident to recommend this program?" The questions were used in the previous studies to assess the acceptability of the internet-delivered program. Open-ended questions will also be used including "How do you think about this program?" "What are the strengths of the program?" "What are the disadvantages of the program?"

ELIGIBILITY:
Inclusion Criteria:

1. Age between 16 to 60;
2. Have a full-time job;
3. Resident of China;
4. Can read and understand Chinese;
5. History with non-cancer pain in past 6 months;
6. Pain score should be at least 2 when using Numeric Rating Scale, a 11-point numeric scale;
7. Own a mobile phone and can access to mobile phone, computer and the internet.

Exclusion Criteria:

1. Hospitalized patients;
2. Experiencing a drug addiction problem;
3. Further medical and surgical treatments or interventions is planned.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-07-05 (Estimated); Study Completion 2020-07-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity and pain interference | Baseline, Week 4, one-month after intervention
  Changes from baseline to Week 4 and one-month after the intervention in pain intensity and pain interference using Brief Pain Inventory

SECONDARY OUTCOMES:
Depression, Anxiety and Stress | Baseline, Week 4, one-month after intervention
  Changes from baseline to Week 4 and one-month after the intervention in depression, anxiety and stress using Depression Anxiety Stress Scale - 21 Scale (DASS-21）. The DASS-21 is a set of three self-reported scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items and divided into subscales. The score of each item ranges feom 0 to 3 (o = do not apply to me at all, 3 = applied to me very much or most of the time). Total score is multiplied by 2 of the sum of each subscales. Higher score indicates the greater degree of the symptom.
Pain self-efficacy | Baseline, Week 4, one-month after intervention
  Changes from baseline to Week 4 and one-month after the intervention in pain self-efficacy using Pain Self-Efficacy Questionnaire (PSEQ). PSEQ is a 10-item questionnaire assessing the confidence people with ongoing pain have in performing activities while in pain. Score of each item ranges from 0 to 6 (0 = not at all confident, 6 = completely confident). A total score is calculated by adding the scores for each item which ranging from 0 to 60. Higher scores reflect stronger self-efficacy beliefs.
Participant's Satisfaction and acceptability to the program | Week 4
  Participants satisfaction and acceptability to the online pain education program will be assessed at post-treatment by several questions, including "do you think this online pain education program useful?" "does it worth your time following the program?" "would you feel confident to recommend this program to others?" Participants are required to answer the questions by "Yes" or "No". Open-ended question "what are the advantages and disadvantages of the program?" will also be asked. These questions have in the previous studies to assess the acceptability and satisfaction to the internet-delivered program.

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Tse, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Tse MYM. An Online Pain Education Program for Working Adults: Pilot Randomized Controlled Trial. J Med Internet Res. 2020 Jan 14;22(1):e15071. doi: 10.2196/15071. PMID 31934865